CLINICAL TRIAL: NCT02192671
Title: Hepatic Resection Versus Radiofrequency Ablation for Patients With Hepatocellular Carcinoma and Portal Hypertension
Brief Title: HR Versus RFA for HCC in Patients With PHT
Acronym: HR-HCC/PHT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Jian-Hong Zhong, Affiliated Tumor Hospital, Guangxi Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRRFA-HCC/PHT; HRRFA-HCC/PHT (Registry Identifier: Jian-Hong Zhong)
Record Dates: First submitted 2014-07-15; First posted 2014-07-17 (Estimated); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Carcinoma, Hepatocellular; Liver Neoplasms; Neoplasms, Glandular and Epithelial
Keywords: hepatocellular carcinoma; radiofrequency ablation; hepatic resection; portal hypertension; Milan criteria; randomized critical trial
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms; Neoplasms, Glandular and Epithelial; Hypertension, Portal | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hepatic resection (Experimental): Adequate remnant liver volume was 30% for HCC patients without cirrhosis, and >50% for HCC patients with chronic hepatitis, cirrhosis, or severe fatty liver.
  Interventions: Procedure: Hepatic Resection
- Radiofrequency ablation (Active Comparator): RFA is performed in less than one week after clinical diagnosis.
  Interventions: Procedure: Radiofrequency Ablation

INTERVENTIONS:
Procedure: Hepatic Resection — Indications for HR are the presence of appropriate residual liver volume determined by volumetric computed tomography.
  Arms: Hepatic resection
Procedure: Radiofrequency Ablation
  Arms: Radiofrequency ablation

SUMMARY:
The purpose of the investigators' study is to prospectively compare the safety and efficacy of hepatic resection to radiofrequency ablation for hepatocellular carcinoma in patients with portal hypertension.

DETAILED DESCRIPTION:
Cirrhosis is common among patients with hepatocellular carcinoma (HCC); in China, for example, it occurs in approximately 80% of HCC patients. Another common comorbidity of HCC is clinically significant portal hypertension (PHT), which occurs in 25-55% of patients with both HCC and cirrhosis. PHT correlates with the severity of cirrhosis, and it can complicate HCC treatment by increasing the risk of perioperative hemorrhage and liver failure.

Hepatic resection (HR) is a widely used radical therapy for HCC. Although HR is often suitable for HCC patients with cirrhosis, it is widely regarded as unsuitable for HCC patients with PHT because of the potential for postoperative hepatic decompensation. In fact, the absence of PHT is the best predictor of excellent HR outcomes. Guidelines of the American and European Associations for the Study of Liver Disease do not recommend HR as an option for HCC patients with PHT. Several studies, however, have reported that HCC patients with and without clinically significant PHT showed similar short- and long-term outcomes after HR. This controversy is important to resolve because more than 25% of cirrhotic patients with HCC also present with PHT.

Actually, official guidelines recommend liver transplatation for patients with HCC and PHT. However, implementation of liver transplantation is restricted by the lack of liver donation and the high cost of the procedure in many countries, especially China. However, as a minimally invasive therapy, radiofrequency ablation (RFA) is a popular treatment modality for patients with HCC within Milan Criteria. Moreover, randomized controlled trials have validated and proposed its clinical usage.

So here, we plan to address the safety and efficacy of HR comparing with RFA for HCC patients with PHT using a population from Guangxi province of China, where the population shows the highest HCC incidence in the world.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* In the HR group, clinical diagnosis of HCC was confirmed by histopathological examination of surgical samples in all patients; in the RFA group, HCC diagnosis was confirmed by two types of clinical imaging (ultrasonography, computed tomography, or magnetic resonance imaging), togetherwith a serum level of α-fetoprotein higher than 400 ng/mL. If diagnosis based on imaging andα-fetoprotein level was uncertain, needle biopsy was performed.
* Tumor stage fitted into Milan Criteria
* Patients with clinically relevant portal hypertension, which is defined as the presence of esophageal varices and/or a platelet count of less than 100 000 per μL in association with splenomegaly.
* Patients have Child-Pugh A or B liver function
* No previous neoadjuvant treatment
* No evidence of metastasis to the lymph nodes and/or distant metastases on the basis of preoperative imaging results and perioperative findings
* No malignancy other than HCC for 5 years prior to the initial HCC treatment

Exclusion Criteria:

* History of cardiac disease
* Known history of human immunodeficiency virus (HIV) infection
* Known Central Nervous System tumors including metastatic brain disease
* History of organ allograft
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* Any condition that is unstable or which could jeopardize the safety of the patient and his/her compliance in the study
* Pregnant or breast-feeding patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-05 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 3 years
Hospital mortality | 90 day

SECONDARY OUTCOMES:
Recurrence rate | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Hepatobilliary Surgery, Affiliated Tumor of Guangxi University, Nanning, Guangxi, China